CLINICAL TRIAL: NCT00090545
Title: A Phase II Study of BAY 43-9006 (Sorafenib) in Metastatic, Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Dahut Jr., M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040262; 04-C-0262; NCT00093431 (obsolete NCT alias)
Record Dates: First submitted 2004-08-27; First posted 2004-08-27 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
Keywords: Hormone-Refractory; Proteomics; Angiogenesis; VEGFR; Prostate Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First Stage - disease progression (Experimental): The first stage was to rule out the probability of 4 month progression free survival.
  Patients were given 400 mg BAY 43-9006 orally twice daily in 28 day cycles.
  Interventions: Drug: BAY 43-9006
- Second Stage - increased accrual (Experimental): Due to prostatic specific antigen and radiographic discordance during the first stage, the protocol was amended to allow accrual to a second stage.
  Patients were given 400 mg BAY 43-9006 orally twice daily in 28 day cycles.
  Interventions: Drug: BAY 43-9006

INTERVENTIONS:
Drug: BAY 43-9006 — 400 mg BAY 43-9006 orally twice daily in 28 day cycles.
  Other Names: sorafenib

SUMMARY:
BAY 43-9006 (Sorafenib) is an experimental cancer drug produced by Bayer Health Care Corporation. It represents a new class of anticancer agents known as bi-aryl ureas. This study will investigate its effect on prostate cancer and its side effects. Researchers expect to enroll a maximum of 46 men with prostate cancer for this study. The duration of the study will depend on its results.

Before beginning to take the drug, patients will be admitted to the hospital for 2 days, have a medical examination and give blood samples, and have a tumor or bone marrow biopsy. On the first day of the study, patients will begin taking the drug as 2 tablets twice daily, morning and evening. Blood will be taken throughout the day to determine the drug's level in the bloodstream.

Patients will be discharged from the hospital on the second day, and will continue to take the drug twice daily until instructed to stop. During each of the first 4 weeks, patients will be required to have their blood pressure checked. At the end of the first 4 weeks, patients will have a physical examination and blood tests, as well as a second tumor or bone marrow biopsy.

After the first 4 weeks, patients will continue with their drug regimen. At the end of each 4-week cycle, patients will have a physical examination and blood tests. Patients will also have x-Rays, computed tomography (CT) scans, and/or magnetic resonance imaging (MRIs) at every other 4-week examination or as required. Patients will be asked to keep a diary recording the time and amount of their medication for this study.

DETAILED DESCRIPTION:
BAY 43-9006 (Sorafenib) is a potent inhibitor of wild-type and mutant b-Raf and c-Raf kinase isoforms in vitro. In addition, this agent also inhibits p38, c-kit, vascular endothelial growth factor receptor 2 (VEGFR-2) and platelet-derived growth factor receptor beta (PDGFR-beta) affecting tumor growth as well as possibly promoting apoptosis by events downstream of c-Raf. At this time, over 500 patients have been treated with this drug with tolerable side effects.

The primary objective of this study is to determine if BAY 43-9006 (Sorafenib) is associated with a 50% 4 month probability of progression free survival in patients with metastatic androgen independent prostate cancer (AIPC) as determined by clinical, radiographic, and prostatic specific antigen (PSA) criteria.

The secondary objective of this study will be demonstration of biologic effect by the drug in the patient and on the tumor (when possible). Correlative studies will be conducted on serially obtained tissue biopsies, bone marrow biopsies, and white blood cell collections. These laboratory correlates will include elucidation of activation of components of the Raf-extracellular-signal regulated kinase (ERK)-methyl ethyl ketone (MEK) and angiogenesis pathways using protein microarray technologies developed by the National Cancer Institute (NCI)/Food and Drug Administration (FDA) clinical proteomics program.

Per Amendment D, a secondary objective of this study will also be to determine the time to progression measured by clinical and radiographic criteria. The 22 patients treated on the first stage of this protocol will be retrospectively evaluated with respect to this secondary endpoint possible. Please refer to the statistics section for further details.

The combination of correlated clinical and laboratory endpoints with emphasis on molecular signaling will provide new information on the anti-tumor effects helping to characterize its role in the treatment of androgen independent prostate cancer (AIPC).

ELIGIBILITY:
* INCLUSION CRITERIA

Patients must have histopathological confirmation of prostate cancer by the Laboratory of Pathology of the National Cancer Institute (NCI) or Pathology Department of the National Naval Medical Center prior to entering this study. Patients whose pathology specimens are no longer available may be enrolled in the trial if the patient has a clinical course consistent with prostate cancer and available documentation from an outside pathology laboratory of the diagnosis. In cases where original tissue blocks or archival biopsy material is available, all efforts should be made to have the material forwarded to the research team for use in correlative studies.

Patients must have metastatic progressive androgen-independent prostate cancer. There must be radiographic evidence of disease after primary treatment with either surgery or radiotherapy that has continued to progress despite hormonal agents. Progression requires that a measurable lesion is expanding, new lesions have appeared, and/or that prostatic specific antigen (PSA) is continuing to rise on successive measurements. Patients on flutamide must have disease progression at least 4 weeks after withdrawal. Patients on bicalutamide or nilutamide must have progression at least 6 weeks after withdrawal.

Patients may have had no more than 1 previous cytoxic chemotherapeutic line.

Because no dosing or adverse event data are currently available on the use of BAY 43-9006 (Sorafenib) in patients less than 18 years of age, children are excluded from this study.

Patients must have a life expectancy of more than 3 months.

Patients must have a performance status of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) criteria.

Patient must have adequate organ function as defined below:

Leukocytes greater than or equal to 3,000/microL

Absolute neutrophil count greater than or equal to 1,500/microL

Platelets greater than or equal to 100,000/microL

Total bilirubin less than or equal to 1.5 X institutional upper limits of normal

Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase(SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 X institutional upper limit of normal

Creatinine less than or equal to 1.5 X institutional upper limits of normal OR:

Creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.

Hormonal profile: all patients who have not undergone bilateral surgical castration must continue suppression of testosterone production by appropriate usage of gonadotropin releasing hormone (GnRH) agonists.

Patients must not have other invasive malignancies (within the past two years with the exception of non-melanoma skin cancers or non-invasive bladder cancer).

Patients must be able to understand and sign an informed consent form.

Concurrent use of bisphosphonates will be allowed for patients with known bone metastases

Patients who require hematopoietic growth factor support (e.g. epogen, darbepoetin), non-steroidal anti-inflammatory drug (NSAIDs), and other maintenance medications prior to study entry will be allowed to continue their supportive therapies.

The effects of BAY 43-9006 (Sorafenib) on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because Raf-kinase inhibitors are known to be teratogenic, men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.

EXCLUSION CRITERIA

Patients who have had chemotherapy or radiotherapy (including radioisotopes) within 4 weeks (6 weeks for nitrosoureas or mitomycin C, greater than 3 months for suramin) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Patients may not be receiving any other investigational agents.

Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006 (Sorafenib)

Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Hypertension as defined by systolic blood pressure in excess of 170 mmHg or diastolic pressure in excess of 100 mmHg. Patients with a history of hypertension that is well controlled on medication will not be excluded. Patients may not be on either verapamil or diltiazem while on study. Use of calcium channel blocker should be discouraged.

Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006 (Sorafenib). Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

History of bleeding diathesis

Patients on therapeutic anticoagulation are at increased risk from bleeding while on BAY 43-9006 (Sorafenib). Prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for prothrombin time (PT), International normalized ratio (INR) or partial thromboplastin time (PTT) are met: PT less than 1.1 x institutional upper limit of normal; INR less than 1.1; PTT within the institutional limits of normal. These requirements will only be made upon those patients on warfarin.

INCLUSION OF WOMEN AND MINORITIES

Men of all races and ethnic groups are eligible for this trial. Women are excluded by the nature of the disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-09-01 (Actual); Primary Completion 2007-09-01 (Actual); Study Completion 2009-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Dahut, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klotz L. Hormone therapy for patients with prostate carcinoma. Cancer. 2000 Jun 15;88(12 Suppl):3009-14. doi: 10.1002/1097-0142(20000615)88:12+3.3.co;2-5. PMID 10898345
- [Background] Peer CJ, Sissung TM, Kim A, Jain L, Woo S, Gardner ER, Kirkland CT, Troutman SM, English BC, Richardson ED, Federspiel J, Venzon D, Dahut W, Kohn E, Kummar S, Yarchoan R, Giaccone G, Widemann B, Figg WD. Sorafenib is an inhibitor of UGT1A1 but is metabolized by UGT1A9: implications of genetic variants on pharmacokinetics and hyperbilirubinemia. Clin Cancer Res. 2012 Apr 1;18(7):2099-107. doi: 10.1158/1078-0432.CCR-11-2484. Epub 2012 Feb 3. PMID 22307138
- [Background] Jain L, Woo S, Gardner ER, Dahut WL, Kohn EC, Kummar S, Mould DR, Giaccone G, Yarchoan R, Venitz J, Figg WD. Population pharmacokinetic analysis of sorafenib in patients with solid tumours. Br J Clin Pharmacol. 2011 Aug;72(2):294-305. doi: 10.1111/j.1365-2125.2011.03963.x. PMID 21392074
- [Background] Jain L, Sissung TM, Danesi R, Kohn EC, Dahut WL, Kummar S, Venzon D, Liewehr D, English BC, Baum CE, Yarchoan R, Giaccone G, Venitz J, Price DK, Figg WD. Hypertension and hand-foot skin reactions related to VEGFR2 genotype and improved clinical outcome following bevacizumab and sorafenib. J Exp Clin Cancer Res. 2010 Jul 14;29(1):95. doi: 10.1186/1756-9966-29-95. PMID 20630084
- [Background] Azad NS, Aragon-Ching JB, Dahut WL, Gutierrez M, Figg WD, Jain L, Steinberg SM, Turner ML, Kohn EC, Kong HH. Hand-foot skin reaction increases with cumulative sorafenib dose and with combination anti-vascular endothelial growth factor therapy. Clin Cancer Res. 2009 Feb 15;15(4):1411-6. doi: 10.1158/1078-0432.CCR-08-1141. PMID 19228742
- [Background] Jain L, Gardner ER, Venitz J, Dahut W, Figg WD. Development of a rapid and sensitive LC-MS/MS assay for the determination of sorafenib in human plasma. J Pharm Biomed Anal. 2008 Jan 22;46(2):362-7. doi: 10.1016/j.jpba.2007.10.027. PMID 18309574
- [Background] Kong HH, Cowen EW, Azad NS, Dahut W, Gutierrez M, Turner ML. Keratoacanthomas associated with sorafenib therapy. J Am Acad Dermatol. 2007 Jan;56(1):171-2. doi: 10.1016/j.jaad.2006.10.032. No abstract available. PMID 17190642
- [Result] Aragon-Ching JB, Jain L, Gulley JL, Arlen PM, Wright JJ, Steinberg SM, Draper D, Venitz J, Jones E, Chen CC, Figg WD, Dahut WL. Final analysis of a phase II trial using sorafenib for metastatic castration-resistant prostate cancer. BJU Int. 2009 Jun;103(12):1636-40. doi: 10.1111/j.1464-410X.2008.08327.x. Epub 2009 Jan 9. PMID 19154507
- [Result] Dahut WL, Scripture C, Posadas E, Jain L, Gulley JL, Arlen PM, Wright JJ, Yu Y, Cao L, Steinberg SM, Aragon-Ching JB, Venitz J, Jones E, Chen CC, Figg WD. A phase II clinical trial of sorafenib in androgen-independent prostate cancer. Clin Cancer Res. 2008 Jan 1;14(1):209-14. doi: 10.1158/1078-0432.CCR-07-1355. PMID 18172272
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2004-C-0262.html

RESULTS

PARTICIPANT FLOW:
Groups:
- First Stage - Disease Progression: The first stage was to rule out the probability of 4 month progression free survival.
  400 mg BAY 43-9006 orally twice daily in 28 day cycles.
- Second Stage - Increased Accrual: Due to prostatic specific antigen and radiographic discordance during the first stage, the protocol was amended to allow accrual to a second stage.
  400 mg BAY 43-9006 orally twice daily in 28 day cycles.
Period: Overall Study
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Started | 22 | 24
Completed | 0 | 0
Not Completed | 22 | 24
Not completed — Disease progression on study | 21 | 17
Not completed — Refused further treatment | 1 | 4
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 9 | 14 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.04) | 68.08 (10.17) | 66.52 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Determine whether BAY 43-9006 when used to treat metastatic prostate cancer is associated with having 50% of Patients Progression Free at 4 Months by clinical, radiographic, and prostatic specific antigen (PSA)criteria.
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 22 | 24
months | 1.83 [1.77 to 3.65] | 3.7 [1.8 to 4.9]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 49 months.
Measure: Count of Participants; unit: Participants
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 22 | 24
Participants | 22 | 23

3. Secondary Outcome: Median Overall Survival
Description: Time from treatment start date until date of death or date last known alive.
Time Frame: Time from treatment start date until date of death or date last known alive, approximately 18.3 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 22 | 24
Months | 18 [1 to 42] | 18.3 [1 to 42]

4. Secondary Outcome: Overall Response Evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Overall response was evaluated by the RECIST. Complete Response (CR) is the disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 2 cycles (1 cycle = 28 days)
Population: For stage 1, not all patients were analyzed for RECIST. Some patients came off study for rising prostatic specific antigen (PSA) only.
Measure: Count of Participants; unit: Participants
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 8 | 24
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1
  Progressive Disease | 8 | 13
  Stable Disease | 0 | 10

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of BAY 43-9006 (Sorafenib)
Description: Plasma concentration-time profile for sorafenib.
Time Frame: 0, 0.25, 0.50, 1, 2, 4, 6, 8, 12, AND 24 hours post dose
Measure: Mean (Full Range); unit: mg/L
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 22 | 24
mg/L | 1.28 [0.88 to 1.87] | 2.57 [1.9 to 3.5]

6. Secondary Outcome: Geometric Mean for Exposure Area Under the Curve (AUC) 0-12
Description: Geometric mean exposure for sorafenib.
Time Frame: 0, 0.25, 0.50, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L.h
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 22 | 24
mg/L.h | 9.76 [6.76 to 14.09] | 18.63 [13.1 to 26.4]

7. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of BAY 43-9006 (Sorafenib)
Description: Time to maximum concentration for sorafenib.
Time Frame: 0, 0.25, 0.50, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
Number analyzed (Participants) | 22 | 24
hours | 0.68 [0.68 to 6.43] | 8 [2 to 12.2]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 49 months.
Arm/Group | First Stage - Disease Progression | Second Stage - Increased Accrual
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/24
Serious Adverse Events (participants affected / at risk) | 2/22 | 6/24
Other Adverse Events (participants affected / at risk) | 22/22 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Stage - Disease Progression (N=22) | Second Stage - Increased Accrual (N=24)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoglobin (Investigations) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 0 (0) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Stage - Disease Progression (N=22) | Second Stage - Increased Accrual (N=24)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 10 (11)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (5) | 11 (13)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (6) | 10 (10)
Alkaline phosphatase (Investigations) | 5 (6) | 7 (7)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 1 (1)
Amylase (Investigations) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 12 (13)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Atrophy, skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Auditory/Ear - Other (Specify,congestion L. ear) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 2 (3) | 3 (4)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 0 (0) | 1 (1)
Conduction abnormality/atrioventricular heart block::AV Block-First degree (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dermatology/Skin - Other (Specify, keratoid canthomas; skin dryness) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (13) | 13 (16)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (7) | 18 (22)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (3)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Gastrointestinal - Other (Specify, soft stool x1 a day) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoglobin (Investigations) | 2 (4) | 7 (8)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Hot flashes/flushes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (5) | 7 (8)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Leukocytes (total WBC) (Investigations) | 0 (0) | 1 (1)
Lipase (Investigations) | 0 (0) | 2 (2)
Lymphopenia (Investigations) | 0 (0) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Mood alteration::Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mood alteration::Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9) | 5 (6)
Neuropathy: sensory (Nervous system disorders) | 3 (3) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 2 (2)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Investigations) | 2 (3) | 1 (1)
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (3)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (4)
Pain::Face (General disorders) | 0 (0) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 0 (0) | 2 (3)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Pain::Kidney (Renal and urinary disorders) | 0 (0) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 1 (1) | 0 (0)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain::Oral-gums (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain::Pain NOS (General disorders) | 0 (0) | 1 (1)
Pain::Pelvis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain::Scrotum (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral arterial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (7) | 10 (11)
Platelets (Investigations) | 0 (0) | 3 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Pulmonary/Upper Respiratory - Other (Specify, phlegm (upper respiratory); upper respiratory)) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (12) | 20 (24)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (5) | 14 (26)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (7) | 3 (4)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 2 (2)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 2 (2)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
Weight loss (Investigations) | 6 (6) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2008-11-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT00090545/Prot_000.pdf